CLINICAL TRIAL: NCT06863870
Title: Assessment of Circulating Tumor Cells and microRNAs in Patients With Metastatic Non-cutaneous Melanoma
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: circMEL 2.0; RC-2022-2773352 (Other Grant/Funding Number: Italian Health Ministry)
Record Dates: First submitted 2025-01-10; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-11

CONDITIONS: Melanoma Neoplasms
Keywords: uveal melanoma; mucosal melanoma; melanoma primary unknown
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the study aims to implement new approaches for the identification of circulating tumor cells and circulating microRNAs, which aim to silence the expression of genes and thus prevent the production of proteins in patients with advanced melanoma (uval, mucosal, of unknown origin). It also aims to verify whether their expression can be related to the prognosis of the disease and the response to treatments.

DETAILED DESCRIPTION:
Here we propose a study to identify a technique for the isolation of circulating tumor cells (CTCs) from blood samples of patients with diagnosis of metastatic melanoma (uveal, mucosal, from primary unknown) to identify a potential role of CTCs and to study the role for circulating microRNAs (miRNAs) in the management of metastatic UM, MM and MUP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UM, MM or MUP
* Diagnosis of metastatic disease
* Age ≥ 18 years, at the time of the tissue collection

Exclusion Criteria:

* Personal medical history of concomitant other cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of metastatic UM or MM or MUP will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Melanoma circulating tumor cell (CTC) count (number of CTC/ml) | At enrollment and at every scheduled follow-up visits throughtout the study (24 months)
  Evaluate CTCs count (number/ml) in patients with metastatic UM, MM and MUP
Circulating microRNAs (copies/ml) | At enrollment and at every scheduled follow-up visits throughtout the study (24 months)
  Evaluate circulating microRNAs expression (copies/ul) in patients with metastatic UM, MM and MUP

SECONDARY OUTCOMES:
Overall Survival (OS) | Throughtout the study duration (24 months) for a minumum of 6 months for each patient
  Evaluate OS throughtout the study period in order to correlate levels of CTC and microRNA with OS of patients with metastatic UM, MM and MUP
To correlate the count of CTC and the expression of circulating microRNAs with patients' prognosis in order to discover liquid biomarkers for prognosis of UM, MM and MUP | Throughtout the study duration (24 months) for a minumum of 6 months for each patient
  Evaluate PFS throughtout the study period in order to correlate levels of CTC and microRNA with PFS of patients with metastatic UM, MM and MUP

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ardizzoni, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No